CLINICAL TRIAL: NCT05722366
Title: Comparison of Acute Responses of Aerobic Exercise and Active Video Games in Coronary Artery Patients
Brief Title: Investigation of Acute Responses of Active Video Games Practice Compared to Exercise in Coronary Artery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Hande Cörüt, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DokuzEU-CAD-001
Record Dates: First submitted 2022-12-19; First posted 2023-02-10 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; active video games; aerobic exercise
MeSH Terms: conditions — Coronary Artery Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Video Game İntervention (Active Comparator): The active video games intervention will be carried out with a virtual reality system (XBOX360, Microsoft, USA) consisting of a console and a sensor.
  Active video games consist of Bowling, River Rush, Rally Ball and Reflex Ridge games.
  Participants will exercise for a total of 25 minutes with light-paced games for warm-up for the first 5 minutes, then brisk games with different body movements until the 15 minutes are complete, and light-paced games for 5 minutes to cool down.
  Participants will complete active video games in the same order.
  Interventions: Other: Active video game
- Aerobic Exercise Intervention (Active Comparator): The exercise intervention will consist of a continuous moderate intensity walking session on the treadmill. After the first 5 minutes of warm-up,a at 55-70% of the peak heart rate reserve(HRR)with a 15-minute walking session, and 5 minutes of cooling down total of 25 minutes of exercise will be performed.
  Interventions: Other: aerobic exercise

INTERVENTIONS:
Other: Active video game — With the closed envelope method, the order in which the participants will perform active video games and aerobic exercise will be determined. It will be applied with 2 weeks between interventions.
  Arms: Active Video Game İntervention
Other: aerobic exercise — With the closed envelope method, the order in which the participants will perform active video games and aerobic exercise will be determined. It will be applied with 2 weeks between interventions.
  Arms: Aerobic Exercise Intervention

SUMMARY:
At least 25 volunteers with a diagnosis of coronary artery disease in the Department of Cardiology of Dokuz Eylul University and who meet the criteria for follow-up and inclusion will participate in the study. Demographic and clinical information of the participants will be questioned. Active video games and exercise sessions will be randomized to last 25 minutes. Before and after the sessions, heart rate, blood pressure, shortness of breath, oxygen saturation and arterial stiffness will be measured. In addition, energy expenditure, heart rate, perceived exertion, shortness of breath and oxygen saturation will be recorded during the sessions. At the end of the sessions, the person will be asked if they enjoy active video games.

DETAILED DESCRIPTION:
Individuals etiology, demographic information (age, gender,marital status, education,occupation),risk factors (smoking,alcohol use,exercise habit),height,weight,curriculum vitae, family history, medications used, and effort test results will be recorded.

Evaluation of energy expenditure: Energy expenditure during active video games and exercise will be evaluated using the activity monitor. The activity monitor will be attached to the upper arm. Its accelerometer measures skin temperature, galvanic skin response and heat flux, as well as energy expenditure during movement.

Evaluation of hemodynamic and pulmonary responses:

Blood pressure: It will be measured with a sphygmomanometer. Perceived effort: The degree of perceived effort will be evaluated with the Modified Borg scale.

Shortness of breath: Shortness of breath will be assessed with the Modified Borg scale.

Heart rate and Oxygen saturation: It will be evaluated by pulse oximetry. Evaluation of vascular responses: Arterial stiffness will be assessed to assess vascular responses to active video games and exercise. Arterial stiffness will be measured with a noninvasive method with the help of the SphygmocorXCEL device, which can automatically measure with the cuff. The patient's age, gender, blood pressure, height, weight, carotid-sternal notch distance between the artery, carotid-femoral artery as the distance between the entered data to the computer after increasing pressure over the brachial artery through a transducer (augmentation index) and again, carotid-femoral pulse wave velocity via the artery (pulse wave velocity) measurements will be made.

The pleasure received from both interventions will be evaluated according to the visual analogue scale (0-10).

Active Video Game Intervention The active video games intervention will be carried out with a virtual reality system (XBOX360, Microsoft, USA) consisting of a console and a sensor.

Active video games consist of Bowling, River Rush, Rally Ball and Reflex Ridge games.

Participants will exercise for a total of 25 minutes with light-paced games for warm-up for the first 5 minutes, then brisk games with different body movements until the 15 minutes are complete, and light-paced games for 5 minutes to cool down.

Participants will complete active video games in the same order. Aerobic Exercise Intervention The exercise intervention will consist of a continuous moderate-intensity walking session on the treadmill. After the first 5 minutes of warm-up, at 55-70% of the peak heart rate reserve(HRR)with a 15-minute walking session, and 5 minutes of cooling down a total of 25 minutes of exercise will be performed.

Blood pressure, heart rate, oxygen saturation, dyspnea, and perceived general fatigue (Mod.Borg 0-10) of the participants will be evaluated before the interventions, at the end of the loading, after the exercise, and 5 minutes after the intervention. Before and after the sessions arterial stiffness will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with coronary artery disease
* Being clinically stable
* Becoming a volunteer

Exclusion Criteria:

* The presence of unstable angina
* The presence of a pacemaker
* The presence of cardiomyopathy
* The presence of a high cardiovascular risk
* The presence of November severe neurological, pulmonary and musculoskeletal system diseases
* The patient wants to quit the study

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Exercise load end heart rate | At the 15th minute of the exercise after the warm-up.
  It will be measured with a pulse oximeter at the end of 15 minutes of exercise loading after warming up.
Exercise load end blood pressure | At the 15th minute of the exercise after the warm-up.
  It will be measured with a sphygmomanometer at the end of 15 minutes of exercise loading after warming up.
Exercise load end perceived effort | At the 15th minute of the exercise after the warm-up.
  The degree of perceived effort will be evaluated with the modified borg scale (M.Borg 0-10)at the end of 15 minutes of exercise loading after warming up. As the modified borg score of the person increases, the perceived effort will increase.
Exercise load end oxygen saturation | At the 15th minute of the exercise after the warm-up.
  Oxygen saturation will be evaluated by pulse oximetry at the end of 15 minutes of exercise loading after warming up.
Exercise load end shortness of breath | At the 15th minute of the exercise after the warm-up.
  Shortness of breath will be assessed with the modified borg scale(M.Borg 0-10) at the end of 15 minutes of exercise loading after warming up.As the modified borg score of the person increases, the perceived shortness of breath will increase.

SECONDARY OUTCOMES:
Evaluation of energy expenditure | ''During exercise intervention, average 25 minutes''
  Energy expenditure during active video games and exercise will be evaluated using the activity monitor. The activity monitor will be attached to the upper arm. Its accelerometer measures skin temperature, galvanic skin response and heat flux, as well as energy expenditure during movement.
Evaluation of Arterial stiffness | Before interventions
  Arterial stiffness will be measured with a noninvasive method with the help of the SphygmocorXCEL device, which can automatically measure with the cuff. By means of a transducer, the pressure on the brachial artery will be increased (augmentation index) and carotid-femoral pulse wave velocity (pulse wave velocity) measurements will be made over the artery.
Evaluation of Arterial stiffness | ''First minutes'' after the intervention
  Arterial stiffness will be measured with a noninvasive method with the help of the SphygmocorXCEL device, which can automatically measure with the cuff. By means of a transducer, the pressure on the brachial artery will be increased (augmentation index) and carotid-femoral pulse wave velocity (pulse wave velocity) measurements will be made over the artery.
Baseline Blood pressure | Before interventions
  Systolic and diastolic blood pressure will be measured with a sphygmomanometer.
End of intervention blood pressure | Within the first minutes after the intervention
  Systolic and diastolic blood pressure will be measured with a sphygmomanometer.
Evaluation blood pressure | 5 minutes after exercises
  Systolic and diastolic blood pressure will be measured with a sphygmomanometer.
Baseline heart rate | Before interventions
  Heart rate will be evaluated by pulse oximetry.
End of intervention heart rate | ''First minutes'' after the intervention
  Heart rate will be evaluated by pulse oximetry.
Evaluation heart rate | 5 minutes after exercises
  Heart rate will be evaluated by pulse oximetry.
Baseline perceived effort | Before interventions
  The degree of perceived effort will be evaluated with the Modified Borg scale(M.Borg 0-10).As the modified borg score of the person increases, the perceived effort will increase.
End of intervention perceived effort | Within the first minutes after the intervention
  The degree of perceived effort will be evaluated with the Modified Borg scale(M.Borg).As the modified borg score of the person increases, the perceived effort will increase.
Evaluation perceived effort | 5 minutes after exercises
  The degree of perceived effort will be evaluated with the Modified Borg scale(M.Borg).As the modified borg score of the person increases, the perceived effort will increase.
Baseline Shortness of breath | Before interventions
  Shortness of breath will be assessed with the Modified Borg scale(M.Borg).As the modified borg score of the person increases, the perceived shortness of breath will increase.
End of intervention Shortness of breath | ''First minutes'' after the intervention
  Shortness of breath will be assessed with the Modified Borg scale(M.Borg).As the modified borg score of the person increases, the perceived shortness of breath will increase.
Evaluation Shortness of breath | 5 minutes after exercises
  Shortness of breath will be assessed with the Modified Borg scale(M.Borg).As the modified borg score of the person increases, the perceived shortness of breath will increase.
Baseline Oxygen saturation | Before interventions
  Oxygen saturation will be evaluated by pulse oximetry.
End of Oxygen saturation | ''First minutes'' after the intervention
  Oxygen saturation will be evaluated by pulse oximetry.
Evaluation Oxygen saturation | 5 minutes after exercises
  Oxygen saturation will be evaluated by pulse oximetry.
Enjoyment of interventions | 5 minutes after interventions
  The enjoyment received from both interventions will be evaluated according to the visual analogue scale (0-10).As the visual analog scale score increases, the person's satisfaction with the exercise increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylül University, Izmir, Balcova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No